CLINICAL TRIAL: NCT01895153
Title: The Efficacy of Pentosan Polysulfate Sodium,Hydrodistension and Combination Therapy in Patients With Bladder Pain Syndrome
Brief Title: Efficacy Study of Pentosan Polysulfate Sodium,Hydrodistension and Combination Therapy for Bladder Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, professor,MD,PhD, Samsung Medical Center
Other Study IDs: 2012-03-029
Record Dates: First submitted 2013-06-07; First posted 2013-07-10 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Bladder Pain Syndrome; Pentosan Polysulfate; Hydrodistension
Keywords: bladder pain syndrome; pentosan polysulfate; hydrodistension
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- pentosan polysulfate cohort: pentosan polysulfate monotherapy
- hydrodistension(HD) cohort: hydrodistension(HD) monotherapy
- combination cohort: combination therapy of pentosan polysulfate and hydrodistension.

SUMMARY:
The efficacy of pentosan polysulfate sodium, hydrodistension and combination therapy in patients with bladder pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. men and women who were over 18 years old and had symptoms over 6 months.
2. 4 or more with an pain visual analogue score
3. 12 or more O'Leary-Sant Intersttial Cystitis questionnaire (IC-Q) symptom and problem score and with a pain score and nocturia score of 2 or more.

Exclusion Criteria:

1. history of hydrodistention,augumentation cystoplasty due to IC/BPS
2. pentosan polysulfate sodium (Elmiron) history over 1 month within 6 months.
3. Women of child-bearing potential who were pregnant or nursing
4. mean voided volume lesser than 40ml or over than 400ml.
5. hematuria exceeds 1+ in the urinary dipstick (dipstick) examination.
6. urinary tract infection during run-in periods.
7. genitourinary tuberculosis or bladder,urethral and prostate cancer
8. recurrent urinary tract infection
9. history of hystrectomy,mid-urethral sling,pelvic organ prolapse repair,vaginal delivery or Cesarean section,prostate opreation or treatment etc within 6months.
10. neurologic disease history of cerebral infaction,multiple sclerosis or parkinsonism etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Bladder pain syndrome patients have not been treated with hydrodistention.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2012-04; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
the change of IC-Q symptom index(ICSI)score from baseline to 6 months after each treatment | 6months

SECONDARY OUTCOMES:
The change of voiding dairy parameters(mean number of micturition,Urgency etc) after each treatment. | 1,2,4 and 6months after each treatment .
The change of O'Leary-Sant Intersttial Cystitis questionnaire (IC-Q)score after each treatment | 1,2,4 and 6months after each treatment .
The change of Pelvic Pain and Urgency/Frequency Patient Symptom Scale (PUF) | 1,2,4 and 6months after each treatment .
The change of Global Response Assessment(GRA) score | 1,2,4 and 6months after each treatment .
The change of EQ-5D Health Questionnaire score | 1,2,4 and 6months after each treatment .
The change of Brief Pain Inventory-short form(BPI-sf) score | 1 and 6months after each treatment.
The estimation of safty and Complications for each treatment | 1,2,4 and 6months after each treatment .

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, MD,Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea